CLINICAL TRIAL: NCT03537118
Title: Routine Ultrasound Guidance for Vascular Access for Cardiac Procedures: a Randomized Trial
Brief Title: Routine Ultrasound Guidance for Vascular Access for Cardiac Procedures
Acronym: UNIVERSAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNIVERSAL.2018
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Myocardial Infarction; Coronary Artery Disease; Myocardial Ischemia
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoroscopic + Ultrasound Guidance (Experimental)
  Interventions: Procedure: Fluoroscopic + Ultrasound Guidance
- Fluoroscopic Guidance Alone (No Intervention)

INTERVENTIONS:
Procedure: Fluoroscopic + Ultrasound Guidance — Fluoroscopic Guidance Alone
  Arms: Fluoroscopic + Ultrasound Guidance

SUMMARY:
A randomized, controlled trial to determine whether the use of ultrasound guidance for vascular access during coronary angiography or percutaneous coronary intervention (PCI) will reduce the rates of major vascular complications.

DETAILED DESCRIPTION:
Patients who will undergo a coronary angiography or PCI using femoral access will be allocated to either: 1) femoral access using fluoroscopic and ultrasound guidance, or 2) femoral access using fluoroscopic guidance alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patient referred for coronary angiography or percutaneous coronary intervention (PCI) in whom femoral access is planned.
2. Planned femoral access

Exclusion Criteria:

1. Age ≤ 18 years
2. STEMI
3. Absence of palpable femoral pulse

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Incidence of major vascular complications | up to 30 days post-procedure
  Femoral artery pseudoaneurysm, AV fistula, retroperitoneal bleed, large hematoma (>5 cm), ischemic limb requiring intervention or surgery, or major bleed based on BARC II, III, or V criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit S Jolly, MD, Principal Investigator — Population Health Research Institute; Tej Sheth, MD, Principal Investigator — Population Health Research Institute; Jose Winter, MD, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Strauss SA, Ma GW, Seo C, Siracuse JJ, Madassery S, Truesdell AG, Pereira K, Korngold EC, Kayssi A. Ultrasound-guided versus anatomic landmark-guided percutaneous femoral artery access. Cochrane Database Syst Rev. 2025 Mar 28;3(3):CD014594. doi: 10.1002/14651858.CD014594.pub2. PMID 40152297
- [Derived] Jolly SS, AlRashidi S, d'Entremont MA, Alansari O, Brochu B, Heenan L, Skuriat E, Tyrwhitt J, Raco M, Tsang M, Valettas N, Velianou JL, Sheth T, Sibbald M, Mehta SR, Pinilla-Echeverri N, Schwalm JD, Natarajan MK, Kelly A, Akl E, Tawadros S, Camargo M, Faidi W, Bauer J, Moxham R, Nkurunziza J, Dutra G, Winter J. Routine Ultrasonography Guidance for Femoral Vascular Access for Cardiac Procedures: The UNIVERSAL Randomized Clinical Trial. JAMA Cardiol. 2022 Nov 1;7(11):1110-1118. doi: 10.1001/jamacardio.2022.3399. PMID 36116089
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140